CLINICAL TRIAL: NCT03283111
Title: Correlation Analysis of T-lymphocyte Subsets and Prognosis in Autologous Stem Cell Transplantation (ASCT) for Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jun Zhu, Principal Investigator, Clinical Professor, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSCO-LWP
Record Dates: First submitted 2017-09-05; First posted 2017-09-14 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- autologous stem cell transplantation (Experimental): Lymphoma patients received autologous stem cell transplantation for the first time
  Interventions: Biological: autologous stem cell transplantation

INTERVENTIONS:
Biological: autologous stem cell transplantation — autologous stem cell transplantation

SUMMARY:
This is a retrospective, single-center, non-randomized, non-controlled study. This study aims to explore the effect of T-lymphocyte subsets changes in immunologic reconstitution and prognosis in lymphoma patients who were treated by autologous stem cell transplantation.

DETAILED DESCRIPTION:
High dose chemotherapy combined with autologous peripheral blood stem cell transplantation is the consolidation treatment for advanced lymphoma patients and approved for treating recurrent and refractory lymphoma by prolonging progression-free survival significantly while also improving quality of life. Evidences to date, have validated that changes of T-lymphocyte subsets after autologous stem cell transplantation associated closely with immunologic reconstitution, and have produced amazing effects in prognosis. Whether T-lymphocyte subsets changes could serve as an effective index for prognosis has been a serious question for lymphoma patients treated by autologous stem cell transplantation. In this study, the investigators explore the changes of T-lymphocyte subsets in lymphoma patients before and after autologous stem cell transplantation, and evaluate the significant effect of T-lymphocyte subsets changes in immunologic reconstitution and prognosis in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women≥18 years, <65 years;
2. Lymphoma patients treated by autologous stem cell transplantation for the first time;
3. ECOG ≤ 2;
4. Ccr ≥ 50 ml/min;
5. ALT, AST and TBIL≤2.5-fold upper normal range;
6. Satisfactory heart and lung function;
7. Women of reproductive potential must have a negative pregnancy test. Male and female of reproductive potential must agree to practice birth control during the study and one year post study;
8. Good compliance and sighed informed consent voluntarily.

Patients should be conformed to all inclusion criteria above.

Exclusion Criteria:

1. Prior autologous/ allogeneic hematopoietic stem cell transplantation for lymphoma;
2. Senior or uncontrolled virus injection: HIV, TP, hepatitis virus;
3. Serious complications;
4. LVEF<55%;
5. Atopy or allergy to biological product derived from colibacillus;
6. Women who are breastfeeding, pregnant or refused to practice contraception;
7. Severe mental or nervous system diseases;
8. Severe abnormalities of heart, lung and central nervous system symptoms;
9. Patients with sickle cell disease, erythronoclastic anemia or other hematological disease which has an impact on medullary hematopoiesis;
10. Enrolled in other study currently or 30 days before screen;
11. Patients, in the opinion of investigators, may not be eligible or are not able to comply with the study.

Patients conformed to any of above criteria should be excluded from this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
  Progression-free survival serves as an effective index to analysis the correlation of T-lymphocyte subsets and prognosis. And it would be measured within 2 years.
Overall survival | 2 years
  The investigators would measure the overall survival of participants within 2 years. Overall survival serves as an effective index to analysis the correlation of T-lymphocyte subsets and prognosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China